CLINICAL TRIAL: NCT01073176
Title: Training Executive, Attention and Motor Skills (TEAMS): Preliminary Studies
Acronym: TEAMS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Queens College, The City University of New York (Other)
Responsible Party: Principal Investigator, Jeffrey Halperin, Distinguished Professor of Psychology, Queens College, The City University of New York
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21MH085898 (NIH)
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Executive function; Preschool children; Treatment; Memory; Attention; Training; Cognitive enhancement
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TEAMS (Experimental): TEAMS has been designed to promote executive skills, memory and fine motor control, and includes game-like activities that allow for increases in task complexity.
  Interventions: Other: TEAMS (Training Attention Executive and Motor Skills)

INTERVENTIONS:
Other: TEAMS (Training Attention Executive and Motor Skills) — Training Executive, Attention and Motor Skills (TEAMS) is a new research program for preschool children with Attention-Deficit/Hyperactivity Disorder (ADHD) that attempts to use game-like activities and physical exercise to promote the growth of neural processes that underlie the core features of the disorder (e.g., hyperactivity, impulsivity) as well as associated areas of difficulty (e.g., socialization, motor skills). These activities are implemented at home and in supervised playgroups at no cost to families and are coupled with extensive parental education about ADHD symptoms and associated impairments.
  Other Names: Cognitive enhancement

SUMMARY:
Training Executive, Attention and Motor Skills (TEAMS) is a new research program for preschool children with Attention-Deficit/Hyperactivity Disorder (ADHD) that attempts to use game-like activities and physical exercise to promote the growth of neural processes that underlie the core features of the disorder (e.g., hyperactivity, impulsivity) as well as associated areas of difficulty (e.g., socialization, motor skills). These activities are implemented at home and in supervised playgroups at no cost to families and are coupled with extensive parental education about ADHD symptoms and associated impairments.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 4.0 and less than 6.0 years of age;
2. Receive a T-score on the Hyperactivity scale of the Behavior Assessment System for Children, Second Edition (BASC-2) of at least 65 (1.5 SD above the mean) by either teacher or parent rating, and a score of at least 60 (1 SD above the mean) by the other rater;
3. Meet diagnostic criteria for ADHD-C or ADHD-HI as ascertained using the Kiddie-SADS, which will be administered to the parent.

Exclusion Criteria:

1. Chronic medical illness or is taking systemic medication;
2. Diagnosed neurological disorder;
3. Full Scale IQ below 80 as measured by the Stanford-Binet - Fifth Edition Abbreviated Battery;
4. Diagnosis of autism, pervasive developmental disorder or post-traumatic stress disorder;
5. Determined to be physically aggressive with other children;
6. Parent enrolled in a parent management training program;
7. Not attending school or day

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Daily Diary of Engagement in Games at Home | Weekly during intervention, 1 month follow-up, 3 month follow-up
  Parents complete diaries indicating the games/exercises that they engaged in with their children, as well as the amount of time per day and the degree to which the activities were enjoyable.

SECONDARY OUTCOMES:
Attention Deficit Hyperactivity Disorder Rating Scale IV(ADHD-RS-IV) | Pre intervention, post intervention, 1 month follow-up, 3 month follow-up
  Parent and teacher ratings of ADHD symptom severity
Parent Satisfaction Questionnaire | Post intervention, 1 month follow-up, 3 month follow-up
  Parents rate the palatability of the intervention across a number of dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Halperin, PhD, Principal Investigator — Queens College, City University of New York
Locations (1):
- Queens College, City University of New York, Flushing, New York, United States